CLINICAL TRIAL: NCT01311635
Title: A Phase I, Open Label, Randomised, 4-way Crossover Study to Investigate the Relative Bioavailability of Single Dose AZD1981 Via 3 Different Tablets in Healthy Men and Healthy Women of Non-childbearing Potential
Brief Title: A Bioavailability Study Comparing 3 Different AZD1981 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist / MD, AstraZeneca R&D
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D9830C00020
Record Dates: First submitted 2011-03-03; First posted 2011-03-09 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Phase 1; bioavailability study; AZD1981; tablets; To study the relative bioavailability of single dose AZD1981 via three different tablets; To compare the bioavailability between three different AZD1981 tablets
MeSH Terms: interventions — AZD1981

ARMS (4):
- Treatment A (Experimental)
  Interventions: Drug: AZD1981, current small-particle tablet
- Treatment B (Experimental)
  Interventions: Drug: AZD1981, new small-particle tablet
- Treatment C (Experimental)
  Interventions: Drug: AZD1981, new small-particle tablet
- Treatment D (Experimental)
  Interventions: Drug: AZD1981, new large-particle table

INTERVENTIONS:
Drug: AZD1981, current small-particle tablet — 3x100 mg per oral, single dose in fasted state
  Arms: Treatment A
Drug: AZD1981, new small-particle tablet — 3x100 mg per oral, single dose
  Arms: Treatment B; Treatment C
Drug: AZD1981, new large-particle table — 3x100 mg per oral, single dose in fasted state
  Arms: Treatment D

SUMMARY:
The purpose of this study is to study the relative bioavailability of AZD1981 when using a new tablet compared to the current tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and postmenopausal or surgically sterile female volunteers aged 18-55, inclusive
* Have a body mass index between 19-30 kg/m2 and weigh at least 50 kg and no more than 100 kg, inclusive
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to screening
* Volunteers must be willing to use barrier methods of contraceptive, unless their partners are post-menopausal, surgically sterile or using accepted contraceptive methods.

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings in the physical examination, clinical chemistry, haematology, urinalysis, vital signs (including body temperature), or ECG assessments at Visit 1, or in vital signs (including body temperature) at Visit 2
* Prolonged QTcF >450 ms or shortened QTcF<340 ms at Visit 1 or family history of long QT syndrome
* History of, or current alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the area under the plasma concentration time-curve from zero to infinity /AUC) and the maximum plasma concentration (Cmax) of AZD1981 | Pharmacokinetic (PK) sampling continuously for 60 h after each single dose, ie day 1-3 for each period.

SECONDARY OUTCOMES:
To evaluate basic systemic PK parameters as follows: | PK sampling continuously for 60 h after each single dose, ie day 1-3 for each period
  * AUC(0-t): area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration
  * tmax: time to reach Cmax
  * t1/2λz: terminal half-life
  * CL/F: apparent plasma clearance
  * MRT: apparent mean residence time
  * Vz/F: apparent volume of distribution during terminal phase
To evaluate the safety and tolerability of AZD1981 by assessment of adverse events, laboratory safety parameters, vital signs, ECG, physical examination and weight | Safety will be monitored continuously and safety assessments will be made on several occasions throughout the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kühn, MD, Principal Investigator — Quintiles AB, Phase 1 Services
Locations (1):
- Research Site, Uppsala, Sweden